CLINICAL TRIAL: NCT00158613
Title: A Prospective, Longitudinal Within-Patient Evaluation of the Effectiveness (Durability) of Carticel® (Autologous Cultured Chondrocytes) Compared to Non-Carticel Surgical Treatment for Articular Cartilage Defects of the Knee.
Brief Title: Study of the Treatment of Articular Repair (STAR)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vericel Corporation (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CARTCEL 012-99
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Articular Cartilage
MeSH Terms: interventions — Drug Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Carticel (autologous cultured chondrocyte) implantation — Each Carticel vial of autologous cultured chondrocytes contains approximately 12 million cells implanted into the defect and secured with a periosteal flap

SUMMARY:
This study is a prospective, longitudinal, multi-center, within patient evaluation of patients with articular cartilage defects of the knee who have had an inadequate response to a prior non-Carticel surgical treatment. Patients who met eligibility criteria were enrolled in the study. Subsequent to implantation with Carticel patients have follow-up every 6-months up to 48-months.

ELIGIBILITY:
Inclusion Criteria:

* Provided written informed consent
* Documented history of at least one Grade III or Grade IV defect (modified Outerbridge classification) on the medial or lateral femoral condyle or trochlea
* Failed prior treatment for articular cartilage defects of the knee, e.g. inadequate response to a non- ACI surgical procedure to treat the lesion, within past 3 yrs
* Patient reported overall knee condition of 5 or less on the Modified Cinn Rating System
* patients must have had a cartilage defect located on the medial or lateral femoral condyle or trochlea which had an inadequate response to a prior arthroscopic or other non-Carticel surgical repair procedure

Exclusion Criteria:

* see above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2000-03; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in the KOOS | Baseline, 6 month, 12 months, 24 months, 36 months, 48 months

SECONDARY OUTCOMES:
Change from Baseline in the Modified Cincinnati Score | 6mo, 12mo, 18mo, 24mo, 30mo, 36mo, 42mo, 48mo
Change from Baseline in the Knee injury and Osteoarthritis Outcome Score (KOOS)Which consists of five sub- categories = Pain, ADL, QOL, Symptoms, Sport | 12mo, 24mo, 36mo, 48mo
Change from Baseline in the SF-36 Health Status Survey | 12mo, 24mo, 36mo, 48mo

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (28):
- United States (25):
  - Kerlan Jobe Orthopaedic Clinic, Los Angeles, California
  - Naval Medical Center San Diego, San Diego, California
  - Santa Monica Orthopedic Group, Santa Monica, California
  - Office of Dr. Noah Weiss, Sonoma, California
  - Denver/Vail Orthopedics, Lone Tree, Colorado
  - University of Connecticut Health Center, Farmington, Connecticut
  - Atlanta Sports Medicine & Orthopaedic Center, Atlanta, Georgia
  - Midwest Orthopedics, Chicago, Illinois
  - Midwest Orthopaedic Center, Peoria, Illinois
  - Orthopaedics Indianapolis, Indianapolis, Indiana
  - Physician's Clinic of Iowa, Cedar Rapids, Iowa
  - Bluegrass Orthopaedics, Lexington, Kentucky
  - National Naval Medical Center, Bethesda, Maryland
  - Washington Orthopedic & Knee Clinic, Clinton, Maryland
  - Children's Hospital, Boston, Massachusetts
  - Pro Sports Orthopedics, Brookline, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Strong Memorial Hospital, University of Rochester, Rochester, New York
  - Keller Army Hospital, West Point, New York
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Beaumont Bone and Joint, Beaumont, Texas
  - Brooke Army Medical Center, Fort Sam, Houston, Texas
  - Naval Medical Center Portsmouth, Portsmouth, Virginia
  - Advanced Orthopedic Center, Richmond, Virginia
  - Northwest Orthopedic Specialists, Spokane, Washington
- Canada (3):
  - Royal Columbian Hospital, New Westminster, British Columbia
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Fowler Kennedy Sports Medicine Clinic, London, Ontario

REFERENCES:
- [Result] Zaslav K, Cole B, Brewster R, DeBerardino T, Farr J, Fowler P, Nissen C; STAR Study Principal Investigators. A prospective study of autologous chondrocyte implantation in patients with failed prior treatment for articular cartilage defect of the knee: results of the Study of the Treatment of Articular Repair (STAR) clinical trial. Am J Sports Med. 2009 Jan;37(1):42-55. doi: 10.1177/0363546508322897. Epub 2008 Oct 16. PMID 18927254